CLINICAL TRIAL: NCT00684463
Title: Study to Evaluate the Efficacy and Safety of Single IV Doses of Onicit® (Palonosetron) 0.25 mg in the Prevention of Acute and Delayed Nausea and Vomiting Associated With Moderate and Highly Emetogenic Chemotherapy in Colombia
Brief Title: Palonosetron in Moderately and Highly Emetogenic Chemotherapy Induced Nausea and Vomiting (Study P04935)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P04935
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Neoplasms; Nausea; Vomiting
Keywords: Antiemetic
MeSH Terms: conditions — Neoplasms; Nausea; Vomiting | interventions — Palonosetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palonosetron (Experimental): 0.25 mg IV single dose, 30 minutes prior to the administration of the major chemotherapeutic agent
  Interventions: Drug: Palonosetron

INTERVENTIONS:
Drug: Palonosetron — 0.25 mg IV single dose, 30 minutes prior to the administration of the major chemotherapeutic agent.
  Other Names: SCH 734291 - Onicit®

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of single IV doses of Onicit® (Palonosetron) 0.25 mg in the prevention of acute and delayed nausea and vomiting associated with moderate and highly emetogenic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older.
* Histological or cytological confirmation of malignant disease.
* Karnofsky index >= 50%
* Naïve to chemotherapy (First Cycle of chemotherapy IV with moderate or high emetic risk administered during Day 1 of the study, according to modification of the classification of Paul Hesketh's schema published on Annals of Oncology 17: 20-28, 2006 (Appendix 3).
* Patients that voluntarily sign the consent form.

Exclusion Criteria:

* Pregnancy or suspected.
* Patients during breast feeding.
* Inability to understand or cooperate with the study procedures.
* Received any investigational drugs within 30 days before study entry.
* Received any drug with potential anti-emetic efficacy within 24 hours prior to the beginning of the treatment
* Seizure disorders requiring anticonvulsant medication.
* Persistent vomiting due to any organic etiology.
* Experienced any vomiting, nausea or retching, in the 24 hours prior to chemotherapy.
* Any systemic disease different to base disease
* Known current or history of drug or alcohol abuse
* Gastric outlet or intestinal obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2007-04-11 (Actual); Primary Completion 2008-02-22 (Actual); Study Completion 2008-02-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients having achieved complete response (CR), defined as no emetic episodes and no rescue medication. | During 24 hours after administration of chemotherapy.

SECONDARY OUTCOMES:
Proportion of patients who achieved a CR and of those who achieved complete control | Days 1 to 5 at different time intervals for each secondary outcome.
Number of emetic episodes | Days 1 to 5 at different time intervals for each secondary outcome.
Time to first emetic episode; time to administration and need for rescue therapy; and to treatment failure time to first emetic episode or administration of rescue medication | Days 1 to 5 at different time intervals for each secondary outcome.

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Snyopsis — http://www.merck.com/clinical-trials/policies-perspectives.html